CLINICAL TRIAL: NCT03387397
Title: Assessing Differential Adherence to Medications and Quality of Life Among People Living With HIV and Comorbidities
Acronym: TEAMH
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-0063
Record Dates: First submitted 2017-12-11; First posted 2018-01-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: HIV Infection Primary
Keywords: Co-morbidities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — HIV-1 RNA viral load and CD4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Medications (LM) cohort: Patients will be assigned to the Lower Medications (LM) cohort group (N=85) if they received a drug regimen of less than five different medications/day during the study period.
- Higher Medications (HM) cohort: Patients will be assigned to the Higher Medications (HM) cohort group (N=85) if they received a drug regimen of more than 5 different chronic medications/day during the study period.

SUMMARY:
The investigators propose to utilize quantitative and qualitative methodology to better understand the impact of multiple drug use (polypharmacy) on medication adherence as well as the driving forces behind differential adherence in people living with HIV (PLWH) with comorbidities. Since the clinical relevance of differential adherence to antiretroviral therapy (ART) medication has already been demonstrated and associated with virologic failure and a more rapid progression to AIDS and death, it is imperative to understand the driving forces behind differential adherence (selective drug taking) and its impact on treatment outcomes in PLWH with comorbidities. To this end, the investigators propose utilizing self-report adherence data and abstracted medical record data including pharmacy refills to assess medication adherence among PLWH with comorbidities. The information gained regarding patients' clinical outcomes as well as patients' reported treatment adherence, quality of life, beliefs about medications, and treatment satisfaction will provide the investigators with a comprehensive picture of what constitutes successful HIV treatment among those PLWH managing multiple medications. This is particularly important as non-successful treatment may result in low patient satisfaction, breach of patient-provider trust and reduced medication adherence.

DETAILED DESCRIPTION:
Primary Endpoints:

Medication adherence: The investigators will assess medication adherence at baseline and at six months using the following measures:

1. Self-reported adherence to ART using the AIDS-ACTG questionnaire will be assessed at baseline and six months. To measure medication adherence to ART the investigators will use the validated AIDS Clinical Trials Group (ACTG) Adherence Questionnaire. This assessment is considered one of the "gold-standard" ART self-reported adherence questionnaires. The questionnaire assesses the number of doses missed per medication per day over a recall period of the previous four days. Mean number of doses missed is calculated for all ART medications over the four days. In addition, the ACTG questionnaire includes secondary assessments of adherence including a general time-frame question regarding the last time the participant missed taking any medications and an assessment of reasons as to why medications were skipped if they were skipped.
2. Medication adherence using pharmacy refills will be assessed at baseline (using the prior 6 months of pharmacy refill data) and at six months post-intervention (to assess the study period pharmacy refill data). Since self-report measures can be biased by inaccurate patient recall or by social desirability, the investigators will also measure medication adherence using pharmacy refill data. Adherence using pharmacy refills has been correlated with a wide range of outcomes for patients with cardiovascular as well as other diseases. To measure medication adherence using pharmacy refills the investigators will use the proportion of days covered (PDC) which is used when multiple medications are used concomitantly. PDC = number of days covered by prescription fills/number of days between the first prescription fills during the measurement period and the end of the measurement period (180 days). The patients' will have two measurement periods: 1) 6 months prior to enrollment and 2) the study period beginning on the date of enrollment (index date) and extending through the last day of the study period (six months) or until the last day of follow-up due to death or disenrollment. It is important to note that PDC calculates the days when the patient is covered for all medications in a regimen for the particular study period. The investigators will assess not only the overall medication adherence, but also adherence to each medication. The research team has access to all Northwell-Vivo pharmacies' refill data as that information is linked to patients' electronic medical records. In addition, Investigators will be able to access other local pharmacy data (including Specialty Pharmacies) as well as mail-order pharmacy data. Moreover, if a patient is admitted to the hospital at any point during the study period and receives medications from hospital supply, the additional medications will be added.

The investigators will measure treatment adherence (compliance) according to International Society for Pharmacoeconomics and Outcomes Research. Medication adherence will be calculated as a compliance rate over the entire study period. Compliance rate (CR) = number of doses taken/number of doses prescribed over the 180 day study period. This can be calculated overall and per medication prescribed. On the basis of self-report and pharmacy refills patients with non- ART medication adherence of 80% and ART medication adherence of >95% will be categorized as adherent. The investigators have chosen a cut-off percentage of >95% for ART medications because it has been shown that drug resistance is most common among patients with a medication adherence rate of <95%. Therefore, PLWH must adhere to their ART regimen at a rate of >95% to avert physiological deterioration due to HIV rebound. Moreover, the 80% cut-off percentage have been used widely in observational and randomized controlled studies on non-ART medication adherence (diabetes and cardiovascular drugs) and these definitions of sub-optimal adherence have been associated with moderate to severe adverse outcomes. Combination tablets will be counted as one medication. Only prescribed medication will be included in the medication adherence calculations. Vitamins and OTC will not be included, but they will be analyzed in secondary analyses (see below).

Secondary Endpoints:

Quality of life (QoL) will be assessed at baseline and six months: The investigators will use the World Health Organization HIV QoL Brief Scale (WHOQOL-HIV BREF) which is a widely used, validated scale to assess QoL indicators that are most relevant to PLWH. It has sound psychometric properties in use with similar populations. The scale consists of 26 items that measure HIV-specific aspects of QoL. It generates four dimensions on 5-point Likert scales including physical health, psychological health, social relationships, and environment.This instrument usually takes less than five minutes to complete. The raw scores on the subscales are converted into transformed scores ranging from 4-20.

Patients' illness-specific symptoms and medication-specific side effects will be assessed at baseline and at six months: The investigators will assess illness-specific symptoms and medication-specific side effects (MSSE using the HIV Symptom Index Questionnaire (HIV-SIQ). HIV-SIQ is a validated instrument that assesses a total of 20 symptoms on a 5-point Likert scale which also assesses symptom severity. Patients will be asked if the symptom is associated with HIV or the other comorbidity or both. If the symptom is attributed to one illness, then the patient will be asked if it is a consequence of the illness or felt to be due to a medication side- effect. The sum of the symptoms attributed to the illness will constitute the ISS, whereas the number or the sum of the symptoms attributed to medication will constitute the MSSE. This information will be collected and analyzed at the end of the study.

Patients' beliefs about medication s will be assessed at baseline only: The investigators will use the Beliefs about Medicines Questionnaire[(BMQ) to assess patients' reasoning behind adherence or non-adherence (e.g., level of fear about not taking medication). The BMQ in the appendix is specific for HIV but it will be adapted to the specific patient' chronic condition(s). Data on patients' beliefs about HIV and comorbidity medications will be collected through a questionnaire consisting of 18 questions with a 5-point Likert response scale, ranging from 1 (strongly agree) to 5 (strongly disagree). Items are altered for other comorbidities and HIV specifically.

Patients' illness perceptions will be assessed at baseline and at six months: The investigators will use the revised version of the Illness Perception Questionnaire (IPQ) to assess patients' own personal beliefs about their illnesses and their treatments, and their emotional responses towards the treatments. The IPQ was originally developed for cancer patients, but it has been revised to accommodate PLWH and other chronic conditions. Patients will complete the questionnaire in response to each of their chronic conditions (including HIV). The IPQ is a 5-point Likert scale questionnaire ranging from 1 (strongly agree) to 5 (strongly disagree).

Patients' pill burden perceptions will be assessed at baseline only: The investigators will query patients regarding their perceptions of pill burden using the Pill Burden Questionnaire (PBQ). The PBQ, developed by Zhou et al.,19 consists of five questions with answers ranging from: 1) strongly agree; 2) disagree; 3) neither agree nor disagree.

Health care utilization (hospitalization rates, urgent care center and ER visits) will be assessed prospectively at baseline and at six months and retrospectively 6 months prior patients' enrollment: The investigators will use the electronic medical record (EMR) system, information from Healthix (the Regional Health Information Organization) and self-report to record hospital utilization (i.e., hospitalization rates, urgent care center and ER visits).

Qualitative Measures:

Focus groups: Two focus groups will be conducted to understand the driving forces behind differential adherence and to understand the impact of number of chronic medications on differential adherence. One focus group will consist of 10 randomly selected patients taking between two and four medications and the other will consist of 10 patients taking at >5 (methodology described below), in order to better understand patient-related as well as non-patient-related factors that could be potentially associated with non-adherence including number of chronic medications. Patient-related factors may include forgetfulness, adherence fatigue, lack of routinization, poor understanding of the relationship between non-adherence and disease progression, depression, anxiety, drug misuse and patient-physician relationship, whereas non-patient-related factors may include environmental factors such as, inconvenience of treatment, insurance-related issues/limitations, poor access to healthcare and medications or medication factors such as complexity of regimen and side effects. The investigators will query as to whether adherence patterns vary by medication and what factors, if any, drive differential adherence such as, fear of consequences of non-adherence, symptom burden, medication side effects, and prioritization of one illness over another. The investigators also will discuss patients' perceptions of pill burden, which may impact medication adherence. The term "pill burden" refers not only to the number of pills that a patient is taking daily, but it is also a function of the difficulty [i.e., pill size, pill form (capsule vs tablet), and method of ingestion (swallow vs chew)] patients have with taking the prescribed doses.

ELIGIBILITY:
Inclusion Criteria

All patients must:

* be HIV infected
* be English speaking
* be 18 years or older
* have at least one comorbidity requiring, at least, one additional chronic medication (defined as a medication that the person needs to be taking for at least six months).
* Receiving care at North Shore University Hospital Center for AIDS Research and Treatment

Exclusion Criteria

* Evidence of cognitive impairment that limits the ability to complete the intervention
* Terminally ill patients will be also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with HIV who have at least one comorbidity and are taking medications for both conditions for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Self-reported adherence to antiretroviral therapy (ART) | baseline and 6 months
  To measure medication adherence to ART the investigators will use the validated AIDS Clinical Trials Group (ACTG) Adherence Questionnaire. This assessment is considered one of the "gold-standard" ART self-reported adherence questionnaires. The questionnaire assesses the number of doses missed per medication per day over a recall period of the previous four days. Mean number of doses missed is calculated for all ART medications over the four days. A higher mean, indicates more doses missed.

SECONDARY OUTCOMES:
Quality of Life (QoL) | Change from baseline QoL at six months
  Quality of life (QoL) will be assessed at baseline and six months: The investigators will use the World Health Organization HIV QoL Brief Scale (WHOQOL-HIV BREF) which is a widely used, validated scale to assess QoL indicators that are most relevant to PLWH. It has sound psychometric properties in use with similar populations. The scale consists of 26 items that measure HIV-specific aspects of QoL. It generates four dimensions on 5-point Likert scales including physical health, psychological health, social relationships, and environment. This instrument usually takes less than five minutes to complete. The raw scores on the subscales are converted into transformed scores ranging from 4-20.
Patients' illness-specific symptoms and medication-specific side effects | Change from patients' baseline illness-specific symptoms and medication-specific side effects at six months
  The investigators will assess illness-specific symptoms and medication-specific side effects (MSSE using the HIV Symptom Index Questionnaire (HIV-SIQ). HIV-SIQ is a validated instrument that assesses a total of 20 symptoms on a 5-point Likert scale which also assesses symptom severity. A greater score indicates greater burden of symptoms.
Patients' beliefs about medication's | Change from patients' baseline beliefs about medication's at six months
  The investigators will use the Beliefs about Medicines Questionnaire (BMQ) to assess patients' reasoning behind adherence or non-adherence. The BMQ comprises two sections: the BMQ-Specific (SpecificNecessity and Specific-Concerns; 10 items), that assesses beliefs about the medication prescribed for personal use, and the BMQ-General (General-Harm and General-Overuse; eight items), which assesses beliefs about medication in general. All items have a five-point Likert answer option, which varies from strongly agree to strongly disagree. Higher scores indicate stronger beliefs about the corresponding concepts in each sub-scale (ie, more negative beliefs about medicines).
Patients' illness perception's | Change from patients' baseline illness perception's at six months
  The investigators will use the revised version of the Illness Perception Questionnaire (IPQ) to assess patients' own personal beliefs about their illnesses and their treatments, and their emotional responses towards the treatments. The IPQ was originally developed for cancer patients, but it has been revised to accommodate PLWH and other chronic conditions. Patients will complete the questionnaire in response to each of their chronic conditions (including HIV). The IPQ is a 5-point Likert scale questionnaire ranging from 1 (strongly agree) to 5 (strongly disagree). A higher schore indicates a more negative perception of a patient's illness.
Patients' pill burden perceptions | Baseline
  The investigators will query patients regarding their perceptions of pill burden using the Pill Burden Questionnaire (PBQ). The PBQ, developed by Zhou et al.,19 consists of five questions with answers ranging from: 1) strongly agree; 2) disagree; 3) neither agree nor disagree. A high score indicates a higher perceived burden.
Hospitalization rates | change from 6 months prior to enrollment up to 6 months post enrollment
  The investigators will use the electronic medical record (EMR) system, information from Healthix (the Regional Health Information Organization) and self-report to record hospital utilization (hospitalization rates). The investigators will use a summed score of number of hospital visits during the study period.
urgent care center rates | change from 6 months prior to enrollment up to 6 months post enrollment
  The investigators will use the electronic medical record (EMR) system, information from Healthix (the Regional Health Information Organization) and self-report to record hospital utilization (urgent care center visits). The investigators will use a summed score of number of urgent care visits during the study period.
Emergency Department visit rates | change from 6 months prior to enrollment up to 6 months post enrollment
  The investigators will use the electronic medical record (EMR) system, information from Healthix (the Regional Health Information Organization) and self-report to record hospital utilization (ED visits). The investigators will use a summed score of number of ED visits during the study period.
HIV viral load | baseline and six months
  To assess the impact of our TEAMH app on medication adherence in PLWH with comorbidities the investigators propose to test HIV Viral Load.
CD4 (cluster of differentiation 4) T-cell counts | baseline and six months
  To assess the impact of our TEAMH app on medication adherence in PLWH with comorbidities the investigators propose to test CD4 T-cell counts.
Medication adherence using pharmacy refills to both ART and non-ART | Change from Medication adherence using pharmacy refills to both ART and non-ART at 6 months
  To measure medication adherence using pharmacy refills the investigators will use the proportion of days covered (PDC). PDC = number of days covered by prescription fills/number of days between the first prescription fills during the measurement period and the end of the measurement period (180 days).

OTHER OUTCOMES:
Qualitative Measures for Focus Group | End of enrollment period ( 6 months)
  Focus Groups -Two focus groups will be conducted to understand the driving forces behind differential adherence and to understand the impact of number of chronic medications on differential adherence. Group 1 will include 10 patients that are in the low medication group taking less than 5 medications. Group 2 will consist of 10 patients taking more than 5 medications (high medication group)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Wallach, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital Division of Infectious Diseases/ Center for AIDS Research and Treatment, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided